CLINICAL TRIAL: NCT00972270
Title: RECOVER II Trial: A Prospective Randomized Trial Investigating the Use of the IMPELLA RECOVER LP 2.5 System in Patients With Acute Myocardial Infarction Induced Hemodynamic Instability
Brief Title: Trial Using Impella LP 2.5 System in Patients With Acute Myocardial Infarction Induced Hemodynamic Instability
Acronym: RECOVER II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study closed due to insufficient enrollment
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Karim Benali, MD/ Chief Medical Officer, Abiomed
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDE: G080021
Record Dates: First submitted 2009-09-02; First posted 2009-09-04 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Arterial Occlusive Disease; Heart Diseases; Myocardial Ischemia; Vascular Disease; Arteriosclerosis; Ischemia
MeSH Terms: conditions — Arterial Occlusive Diseases; Heart Diseases; Myocardial Ischemia; Vascular Diseases; Arteriosclerosis; Ischemia | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMPELLA LP 2.5 (Experimental)
  Interventions: Device: Impella LP 2.5
- Intra-Aortic Balloon Pump (Active Comparator)
  Interventions: Device: Intra-Aortic Balloon Pump

INTERVENTIONS:
Device: Impella LP 2.5 — Insertion of the LP 2.5 IMPELLA circulatory support system that can be placed across the aortic valve using a single femoral site. The device pumps blood from the left ventricle into the ascending aorta at 2.5L/min.
  Arms: IMPELLA LP 2.5
Device: Intra-Aortic Balloon Pump — The Intra-Aortic Balloon Pump consists of a cylindrical balloon that sits in the aorta and counterpulsates.
  Arms: Intra-Aortic Balloon Pump

SUMMARY:
This is a randomized trial investigating the use of the IMPELLA RECOVER LP 2.5 compared to Intra-aortic balloon pump (IABP) in patients with Acute Myocardial Infarction.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Subject presenting with STEMI undergoing primary PCI
* Patient presents with at least 1 of the following:
* Unstable blood pressure
* Tachycardia and tissue hypoperfusion
* The need for intravenous pressor or inotropic support
* Patient presents with STEMI:
* CK-MB>2x normal

Exclusion Criteria:

* Unwitnessed cardiac arrest
* Abnormalities of the aorta
* Recent stroke or TIA
* Mural thrombus in the left ventricle

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Composite rate of major adverse events within 30 days or hospital discharge. | 30 days or discharge
  Composite rate of major adverse events within 30 days or hospital discharge.

SECONDARY OUTCOMES:
Maximum CPO increase from baseline. | Treatment
  Maximum CPO increase from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: William O'Neill, M.D., Principal Investigator — Not affiliated with Abiomed
Locations (11):
- United States (11):
  - Hartford Hospital, Hartford, Connecticut
  - University of Chicago Medical Center, Chicago, Illinois
  - Shawnee Mission, Shawnee Mission, Kansas
  - Valley Hospital, Hawthorne, New Jersey
  - Ohio State University, Columbus, Ohio
  - Riverside Methodist, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Health, Wormleysburg, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah